CLINICAL TRIAL: NCT05411172
Title: The Effect of Chemical Biological Radiological and Nuclear Training Program Based on Mastery Learning Model on the Learning Outcome of Student Nurses
Brief Title: Evaluation of a Model-Based CBRN Training Program
Acronym: CBRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Derya Aslan Huyar, Principal Investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 982d71uk
Record Dates: First submitted 2021-12-16; First posted 2022-06-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chemical Accident; Radiation Exposure; Biological Substance Poisoning
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The Effect of the Education Based on the Mastery Learning Model on the Practical Skills of Student Nurses in Chemical, Biological, Radiological, and Nuclear Hazards.
  The MLM-CBRN Education Program was carried out with the students in the experimental group face-to-face as theoretical and practical education once a week for four weeks.
  Interventions: Behavioral: Mastery Learning Model for Chemical, Biological, Radiological, and Nuclear threats and hazards (MLM-CBRN Education Program) on student nurses
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Mastery Learning Model for Chemical, Biological, Radiological, and Nuclear threats and hazards (MLM-CBRN Education Program) on student nurses — The MLM-CBRN Education Program was carried out with the students in the experimental group face-to-face as theoretical and practical education once a week for four weeks. . The data were collected before and right after the intervention and in the 1st and 3rd months after the intervention using the "Personal Information Form," "Nursing Student CBRN Knowledge Test," "Nursing Student CBRN Attitude Scale," and "Nursing Student CBRN Self-Efficacy Scale." Moreover, only the knowledge scores of the students in the experimental group were collected using the unit follow-up tests, which enabled us to check whether the "Learning Objective" related to the unit taught was achieved. During the skill training, the "START Triage and JumpSTART Triage Skill Check List," Gas Mask Wearing-Removing Skill Check List, and Level C Clothes Wearing-Removing Skill Check List were scored for each student in the experimental group after observing the students twice.
  Arms: Experimental

SUMMARY:
The aim of the study is to evaluate the effect of the Education Program based on the Mastery Learning Model for Chemical, Biological, Radiological, and Nuclear threats and hazards (MLM-CBRN Education Program) on student nurses' knowledge, attitude, self-efficacy, and skill development in chemical, biological, radiological and nuclear threats and hazards. The complete experimental design type was used in the study.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of the Education Program based on the Mastery Learning Model for Chemical, Biological, Radiological, and Nuclear threats and hazards (MLM-CBRN Education Program) on student nurses' knowledge, attitude, self-efficacy, and skill development in chemical, biological, radiological and nuclear threats and hazards. The complete experimental design type was used in the study. The study sample comprised 104 4th-year nursing students (52 in the experimental group, 52 in the control group). The MLM-CBRN Education Program was carried out with the students in the experimental group face-to-face as theoretical and practical education once a week for four weeks. As a criterion for starting a new unit, 80% of the participants needed to receive minimum 70 points from the unit follow-up tests in line with the "Learning Objective" determined within the scope of the Mastery Learning Model. The data were collected before and right after the intervention and in the 1st and 3rd months after the intervention using the "Personal Information Form," "Nursing Student CBRN Knowledge Test," "Nursing Student CBRN Attitude Scale," and "Nursing Student CBRN Self-Efficacy Scale." Moreover, only the knowledge scores of the students in the experimental group were collected using the unit follow-up tests, which enabled us to check whether the "Learning Objective" related to the unit taught was achieved. During the skill training, the "START Triage and JumpSTART Triage Skill Check List," Gas Mask Wearing-Removing Skill Check List, and Level C Clothes Wearing-Removing Skill Check List were scored for each student in the experimental group after observing the students twice.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior nursing undergraduate student
* Not having received CBRN training

Exclusion Criteria:

* Be a full-time worker in a healthcare institution
* Having taken courses on disaster and CBRN

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Individual Information Form | up to 24 weeks
  It consists of items questioning the students' demographic data, their school success, and whether they have received a CBRN education or not.

SECONDARY OUTCOMES:
Nursing Student CBRN Knowledge Test | up to 24 weeks
  Knowledge Test used to determine the knowledge level of nursing students about CBRN consists of 31 items. The answer options of true and false statements. The score that can be obtained from the test varies between 0-31. The results get improve as the points are received.KR-20 was calculated as 0.82

OTHER OUTCOMES:
Nursing Student CBRN Attitude Scale | up to 24 weeks
  To determine their attitudes about kbrn used it.Attitude Scale. The scale consists of 3 sub-factors. Individual attitude (factor 1), professional attitude (factor 2), and social attitude (factor 3). Scores related to the scale score and sub-dimensions are obtained by adding the scores given to the items and dividing them by the number of items. It is a Likert-type scale and is graded between "5" completely agree and "1" strongly disagree. The Cronbach Alpha is 0.92. The score that can be obtained from the test varies between 1-5. The results get improve as the points are received.
Nursing Student CBRN Self-Efficacy Scale | up to 24 weeks
  To determine their self-efficacy about kbrn used it. The Self-Efficacy Scale score is obtained by adding the scores given to the items and dividing them by the number of items. The CBRN attitude scale was grouped under a single factor structure. The scale consists of 9 items. Scores from the scale range from 1 to 5. It is a Likert-type scale. The Cronbach Alpha is 0.90. The score that can be obtained from the test varies between 1-5. The results get improve as the points are received.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Nihal Esin, Study Director — mnesin@istanbul.edu.tr
Locations (1):
- Bursa Uludağ Üniversitesi, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
if requested; training plan, data collection forms used, presentation content used, checklists used, unit follow-up tests used, and case examples used can be shared.
Supporting Information: Study Protocol, ICF
Time Frame: 1-12 months
Access Criteria: have ethics committee approval, Researchers who want to do meta-analysis or systematic review